#### The GlaxoSmithKline group of companies

| Division | ivision : Worldwide Development | |
|---|---|---|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for An open-label extension to Study 200952 in Subjects with Type 2 Diabetes Mellitus to Assess the Long-term Safety and Tolerability of Albiglutide Liquid Drug Product |
|---|---|---|
| Compound Number | : | GSK716155 |
| <b>Effective Date</b> | : | 06-MAR-2017 |

### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 204682.
- This RAP is intended to describe the safety analyses required for the study.
- The study is terminated early with a limited number of subjects (N=8) enrolled and limited data collected (only available at Early Withdrawal and Follow-up visits except one subject had Week 30 visit). Therefore a synoptic CSR is planned and a brief RAP document is prepared accordingly.
- This RAP will be provided to the study team members to convey the content of the content of the final Statistical Analysis Complete (SAC) Deliverable.

#### **Author's Name and Functional Area:**

| PPD | | PPD | | 06-MAR-2017 |
|---|---|---|---|---|
| Senior Bios | tatistician, PPD | Biostatistics Team | Lead, PPD | 00-WAK-2017 |

#### Approved by:

| PPD | | |
|---|---|---|
| 1 | n, Clinical Statistics, R&D Projects Clinical es, GlaxoSmithKline | 06-MAR-2017 |

Copyright 2017 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

### **TABLE OF CONTENTS**

204682

| | | | | PAGE |
|---|---|---|---|---|
| 1. | REPO | RTING & | ANALYSIS PLAN SYNPOSIS | 4 |
| 2. | SUMN<br>2.1.<br>2.2.<br>2.3. | Changes<br>Study Of | | 5<br>6<br>6 |
| 3. | PLAN<br>3.1.<br>3.2. | Interim A | LYSES<br>Analysesalyses | 8 |
| 4. | ANAL' | YSIS POF | PULATIONS | 9 |
| 5. | | | ONS FOR DATA ANALYSES AND DATA HANDLING | 10 |
| 6. | STUD<br>6.1.<br>6.2.<br>6.3.<br>6.4. | Overviev<br>Demogra<br>Exposure | ATION ANALYSES | 11<br>11<br>11 |
| 7. | SAFE 7.1. 7.2. 7.3. 7.4. 7.5. 7.6. | Overview<br>Adverse<br>Clinical L<br>7.3.1.<br>Vital Sign<br>Electroca | OLERABILITY ANALYSES w of Planned Analyses Events aboratory Evaluations Chemistry, Hematology and Urinalysis ns ardiograms genicity | 12<br>13<br>13<br>13 |
| 8. | OTHE | R STATIS | STICAL ANALYSES | 15 |
| 9. | REFE | RENCES. | | 16 |
| 10. | <ul><li>10.1.</li><li>10.2.</li><li>10.3.</li><li>10.4.</li></ul> | Appendix<br>10.1.1.<br>Appendix<br>10.2.1.<br>10.2.2.<br>Appendix<br>10.3.1.<br>Appendix | x 1: Time & Events | |
| | 10.5. | Appendix | x 5: List of Data Displays | <mark>27</mark> |

# 2017N316448\_00

### CONFIDENTIAL

| | | 204682 |
|---------|-------------------------|-----------------|
| 10.5.1. | Data Display Numbering | <mark>27</mark> |
| | Study Population Tables | |
| 10.5.3. | Listings | 28 |
| | 3 | |

204682

# 1. REPORTING & ANALYSIS PLAN SYNPOSIS

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | This study will evaluate the long-term safety, tolerability and pharmacodynamics of albiglutide liquid drug product in subjects with type 2 diabetes mellitus (T2DM) who have completed Study 200952 and satisfy all inclusion/exclusion criteria to enter Study 204682. |
| Protocol | This RAP is based on the protocol (Dated: 28/OCT/2015) of study GSK204682 (GlaxoSmithKline Document Number. : 2015N235104_00] and eCRF Version 2. |
| Primary<br>Objective | To evaluate extended safety, tolerability and immunogenicity data of albiglutide liquid product. |
| Primary<br>Endpoint | AEs and SAEs, clinical laboratory evaluations, physical examinations, vital signs and ECGs |
| | Anti-albiglutide antibody production over time |
| Study<br>Design | This is a 26 week, open-label, single group, multicenter, extension study to Study 200952. This extension study will provide extended safety, tolerability and immunogenicity for the albiglutide liquid drug product. |
| | The extension study will recruit subjects who have completed Study 200952 and satisfy all inclusion/exclusion criteria. Subjects will continue on their current regimen of diet and exercise or stable dose of background metformin (if applicable). |
| | This extension study will comprise 2 study periods: treatment (26 weeks) and post-treatment follow-up (8 weeks). |
| | While at the time the RAP is being prepared, the study is terminated early with a limited number of subjects enrolled. |
| | All subjects will receive 50 mg albiglutide liquid drug product via auto-injector. |
| Analysis<br>Populations | Safety Population |

204682

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

The statistical analysis plan will be done on a limited number of subjects and data (not the full 26 weeks as planned) due to early termination. Only summary for demography and listings for key safety data and immunogenicity will be provided.

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To evaluate extended safety,<br>tolerability and immunogenicity<br>data of albiglutide liquid product. | <ul> <li>AEs and SAEs, clinical laboratory evaluations, physical examinations, vital signs and ECGs</li> <li>Anti-albiglutide antibody production over time</li> </ul> |

### 2.3. Study Design

### 2.3.1. Overview of Study Design and Key Features



Due to early termination the entirety of the study conduct was not carried out.

#### 2.3.2. Study Design

This is a 26 week, open-label, single group, multicenter, extension study to Study 200952. This extension study will provide extended safety, tolerability and immunogenicity of albiglutide liquid drug product.

This study will comprise 2 study periods: treatment (26 weeks) and post-treatment follow-up period (8 weeks).

204682

The extension study will recruit subjects who have completed Study 200952 and satisfy all inclusion/exclusion criteria. Subjects will continue on their current regimen of diet and exercise or stable dose of background metformin (if applicable).

Study treatment will be administered once weekly by s.c. injection in the abdomen, thigh, or upper arm. Subjects will receive 50 mg albiglutide liquid drug product via auto-injector for 26 weeks. The first dose of study treatment will be administered by the subject during the clinic visit (Visit 1, week 26) with supervision from clinic staff. All further doses of study treatment will be self-administered by the subject.

At the time the RAP is being prepared, the study is terminated early with a limited number of subjects enrolled.

204682

# 3. PLANNED ANALYSES

# 3.1. Interim Analyses

No interim analysis is planned for this study.

# 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following step:

All required database cleaning activities have been completed and final database release and database freeze has been declared.

204682

# 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Safety | Comprise of all enrolled subjects who receive<br>at least one dose of study treatment. | Safety |
| | <ul> <li>This population will be analysed according to<br/>the treatment the subject actually received.</li> </ul> | |

# NOTES:

• Please refer to Appendix 5 List of Data Displays which details the population to be used for each displays being generated.

204682

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|--------------|-----------------------------------------------------|
| Section 10.1 | Appendix 1: Time & Events |
| Section 10.2 | Appendix 2: Assessment Windows |
| Section 10.3 | Appendix 3: Values of Potential Clinical Importance |
| Section 10.4 | Appendix 4: Abbreviations and Trademarks |
| Section 10.5 | Appendix 5: List of Data Displays |

### 6. STUDY POPULATION ANALYSES

### 6.1. Overview of Planned Analyses

Table 2 Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 5: List of Data Displays.

Table 2 Overview of Planned Study Population Analyses

| Display Type | Data Display's Generated | | |
|---|---|---|---|
| | Figure | Table | Listing |
| Demography and Baseline Characteristics | | | |
| Demographics and Baseline Characteristics | | Y | Υ |
| Race & Racial Combinations | | | Υ |
| Medical Condition & Concomitant Medications | | | |
| Concomitant Medication | | | Y |
| Exposure | | • | |
| Exposure to Study Drug | | | Υ |

Note: additional tables, listings and figures will be provided in Appendix 5: List of Data Displays.

Following review of the data, additional analyses maybe conducted to further support the evaluation and interpretation of the data.

# 6.2. Demographic and Baseline Characteristics

Demographic and baseline characteristics will be based on the data from the main study 200952 as this is an extension study.

Continuous variables such as age, body mass index, weight, and height will be summarized using descriptive statistics(n, mean, standard deviation, and median, minimum, maximum). Categorical variables including sex and ethnicity will be summarized using numbers and percentages.

Continuous variables such as age, body mass index, weight, and height will be presented in a by-subject listing. Listings will be presented using the safety population, if appropriate and based on the data from the main study 200952.

# 6.3. Exposure to Study Drug

A by-subject listing of study drug administration will also be presented. Overall study drug administration and treatment compliance will be present with the exposure to study drug listing.

<sup>•</sup> Y = Yes display generated.

#### 6.4. Medications

Any medication used during the study will be recorded, which will be updated whenever available throughout the life of the study.

All medications will be listed.

#### 7. SAFETY AND TOLERABILITY ANALYSES

### 7.1. Overview of Planned Analyses

The safety analyses will be based on the safety population.

Table 3 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 5: List of Data Displays.

Table 3 Overview of Planned Safety Analyses

| | Observed | | | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|
| Endpoints | Summary | | Individual | | Summary | | Individual | |
| | Т | F | F | L | Т | F | F | L |
| Adverse Events | | | | Υ | | | | |
| Clinical Laboratory | | | | Υ | | | | |
| Vital Signs | | | | Υ | | | | |
| Electrocardiogram (ECG) | | | | Υ | | | | |
| Immunogenicity | | | | Υ | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

Following review of the data, additional analyses maybe conducted to further support the evaluation and interpretation of the data.

#### 7.2. Adverse Events

All AEs will be coded using MedDRA which will be updated whenever available throughout the life of the study.

All AEs will be listed in a subject data listing.

204682

# 7.3. Clinical Laboratory Evaluations

### 7.3.1. Chemistry, Hematology and Urinalysis

Laboratory parameters include the following tests: hematology, chemistry and urinalysis. Established or generally acknowledged methods, normal ranges, and quality control procedures will be supplied by central lab for the study records.

Hematology parameters include complete blood count with red blood cell indices, white blood cell count with differential, and platelet count. Chemistry parameters (including lipids) include blood urea nitrogen (BUN), potassium, aspartate aminotransferase (AST), total and direct bilirubin, creatinine, sodium, ALT, total protein, calcium, chloride, alkaline phosphatase (ALP), albumin, bicarbonate, uric acid, gamma glutamyl transferase (GGT), estimated glomerular filtration rate (eGFR), and lipids (including total cholesterol, LDL-C, HDL C, triglycerides, free fatty acids). Urinalysis parameters include specific gravity, pH, glucose, protein, blood and ketones by dipstick and microscopic examination (if blood or protein is abnormal).

All laboratory parameters as collected will be presented in by-subject listings at every scheduled assessment time point from Study 200682 and also Week 26 from Study 200952. All listings will be done for the safety population and all laboratory data will be listed including other laboratory tests, such as HIV, Lipase, Amylase, hepatitis B, hepatitis C, TSH, and urine pregnancy test results.

Additionally, the number of subjects with laboratory values of potential clinical concern will be provided in a listing by treatment group and scheduled assessment time point for hematology and chemistry. The criteria for laboratory values of potential clinical concern are detailed in Appendix 3: Values of Potential Clinical Importance.

A listing of laboratory values of potential clinical concern will be provided for liver function tests, including ALT, AST, and total bilirubin. The criteria for liver function tests of potential clinical concern are detailed in Appendix 3: Values of Potential Clinical Importance.

# 7.4. Vital Signs

The vital sign analysis will include systolic blood pressure (mmHg), diastolic blood pressure (mmHg), and heart rate (bpm).

Each vital sign parameter at every scheduled assessment time point will be presented in by-subject listings.

All listings will be produced for the safety population.

204682

# 7.5. Electrocardiograms

ECG parameters collected at each scheduled assessment time point include heart rate, QRS interval, QT interval – Bazett correction (QTcB) (if applicable), QT interval – Fridericia correction (QTcF), RR interval and PR interval.

Each ECG parameter at each scheduled assessment time point will be presented in bysubject listings. All listings will be produced for the safety population.

# 7.6. Immunogenicity

The immunogenicity data will be listed. Immunogenicity listings will be generated only after the unblinding of Study 200952.

204682

# 8. OTHER STATISTICAL ANALYSES

Not applicable.

204682

# 9. REFERENCES

GlaxoSmithKline Document Number 2015N235104\_00. Protocol 204682: An Openlabel Extension to Study 200952 to Evaluate the Long-term Safety, Tolerability and Pharmacodynamics of Albiglutide Liquid Drug Product in Subjects with Type 2 Diabetes Mellitus (28-OCT-2015)

204682

# 10. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 5 | RAP Section 5 : General Considerations for Data Analyses & Data Handling Conventions |
| Section 10.1 | Appendix 1: Time & Events |
| Section 10.2 | Appendix 2: Assessment Windows |
| Section 10.3 | Appendix 3: Values of Potential Clinical Importance |
| Section 10.4 | Appendix 4: Abbreviations and Trademarks |
| Section 10.5 | Appendix 5: List of Data Displays |

# 10.1. Appendix 1: Time & Events

#### 10.1.1. Protocol Defined Time & Events

| | | Treatment | | | | 11End of<br>Treatment | Follow-up <sup>12</sup> | |
|---|---|---|---|---|---|---|---|---|
| Procedure | Extension Study Visit | 1 | 2 | 3 | 4 | 5 | 6 | 7<br>60 |
| | Study Week | 2613 | 30 | 36 | 42 | 48 | 52 | |
| Informed consent for St | udy 204682 | X | | | | Ĭ. | | Ĭ. |
| Inclusion/exclusion crite | ria review <sup>1</sup> | X | | | | | | |
| Full (F) or brief (B) phys | ical exam <sup>2</sup> | F | В | В | В | В | F | F |
| Weight | | X | X | X | X | X | X | X |
| 12-lead ECG <sup>3</sup> | | X | | | | | X | X |
| Vital signs | | X | X | X | X | X | X | X |
| Serum (S)/Urine (U) pregnancy test (WCBP) | | S | U | U | U | Ü | S | |
| Clinical chemistry/hema | X | X | X | | X | X | X | |
| Lipids (including total cholesterol, LDL-C, HDL C, triglycerides, FFAs) <sup>4</sup> | | X | | | | | x | X |
| Urinalysis <sup>5</sup> | | X | | | | | X | |
| HbA <sub>1c</sub> 6,7 | | X | X | X | X | X | X | X |
| FPG 7 | | X | X | X | X | X | X | X |
| eGFR | 7.2 | X | | X | | X | | |
| Immunogenicity sample | 8 | X | X | X | | | X | X |
| Review AE/SAE, concomitant medication and hypoglycemia events | | x | X | x | Х | Х | х | X |
| Advice on diet and exercise9 | | X | X | X | X | X | X | |
| Subject Experience / Satisfaction Exit Questionairre | | | | | | | X | |
| Study treatment dispen | sed | X | X | X | X | X | : | |
| Study treatment compliance <sup>10</sup> | | | X | X | X | X | X | |

WCBP: Women of child bearing potential; FFA: free fatty acids; LDL-c: low density lipoproteins cholesterol; HDL-c: high density lipoproteins cholesterol

- 1. **Before dosing**, the investigator must review **all** inclusion and exclusion criteria to confirm subject's eligibility. If a subject no longer meets all of the eligibility criteria (e.g., there is evidence of a new myocardial infarction (MI) on an ECG or ALT, etc. are out of range), **do not administer the study treatment** and contact the medical monitor to discuss how to proceed (e.g., to determine if repeat testing is warranted).
- 2. Details of full and brief physical examinations are provided in Protocol Section 7.3.3.
- 3. 12-lead ECGs will be obtained **before** measurement of vital signs and collection of blood samples for laboratory testing. See Protocol Section 7.3.5.
- 4. Clinical chemistry and hematology assessments are described in Protocol Section 7.3.6.
- 5. Urine samples should be collected in the early morning.
- 6. Blood samples for HbA<sub>1c</sub> should be collected before administration of study treatment.
- 7. Subjects will have their FPG and HbA<sub>1c</sub> levels evaluated to monitor for potential hyperglycemia.

- 8. Blood samples for immunogenicity are to be collected **before** study drug administration.
- 9. Standard diabetic dietary and exercise advice will be reinforced through the end-of-treatment visit.
- 10. Compliance will be assessed as described in Protocol Section 6.7.
- 11. Subjects who discontinue study treatment should be handled as described in Protocol Section 5.4.
- 12. Follow-up visit for subjects who have discontinued study treatment (see Protocol Section 5.4), or subjects who have completed the 52 week treatment period.
- 13. Visit 1of 204682 is also the end of treatment visit in Study 200952.
- 14. Visit 1 of Study 204682; albiglutide liquid drug product administered to all study subjects.

204682

# 10.2. Appendix 2: Assessment Windows

# 10.2.1. Definitions of Study Day

When study day is used for display or in comparisons the following algorithm will be used:

- Study day = date of assessment date of first dose + 1, if dose of assessment >= first dose date
- Study day = date of assessment date of first dose, if dose of assessment < first dose date

•

Note that the date of first dose is Day 1 and the day before the date of first dose is Day -1 (there is no Day 0).

### 10.2.2. Visit Slotting Algorithm

For all safety parameters to be summarized by visit, nominal visits recorded on the eCRF will be used for the summaries. No visit slotting algorithm will be applied.

204682

# 10.3. Appendix 3: Values of Potential Clinical Importance

# 10.3.1. Laboratory

| | Hematology | | |
|---|---|---|---|
| Laboratory<br>Test | Units | Change from Baseline of<br>Potential Clinical Concern | Potential Clinical Concern<br>Value |
| Basophils | GI/L | None | None |
| Eosinophils | GI/L | None | None |
| Hematocrit | 1 | >0.1 decrease | >0.05 below LLN<br>>0.04 above ULN |
| Hemoglobin | g/L | >25 g/L decrease | >20 g/L below LLN<br>>10 g/L above ULN |
| Lymphocytes | GI/L | None | <0.5 x LLN |
| Monocytes | GI/L | None | None |
| Neutrophils | GI/L | None | <1 GI/L |
| Neutrophil<br>Bands | GI/L | None | None |
| Platelets | GI/L | None | <80 GI/L<br>>500 GI/L |
| Red Blood Cell<br>Count | TI/L | None | None |
| Segmented<br>Neutrophils | GI/L | None | <0.5 x LLN |
| White Blood Cell<br>Count | GI/L | None | >1 GI/L below LLN<br>>5 GI/L above ULN |

| | Chemistry | | |
|---|---|---|---|
| Laboratory<br>Test | Units | Change from Baseline of Potential Clinical Concern | Potential Clinical Concern<br>Value |
| Albumin | g/L | None | >5 g/L above ULN or below LLN |
| Alkaline<br>Phosphatase | U/L | None | >3 x ULN |
| ALT | U/L | None | >3 x ULN |
| AST | U/L | None | >3 x ULN |
| Bicarbonate<br>(Carbon Dioxide<br>Content) | mmol/L | None | <16 mmol/L<br>> 40 mmol/L |
| Blood Urea<br>Nitrogen | mmol/L | None | >2 x ULN |
| Calcitonin | pmol/L | None | >100 |

204682

| | Chemistry | | |
|---|---|---|---|
| Laboratory<br>Test | Units | Change from Baseline of Potential Clinical Concern | Potential Clinical Concern<br>Value |
| Calcium | mmol/L | None | <1.8 mmol/L<br>>3.0 mmol/L |
| Chloride | mmol/L | None | None |
| Creatinine | umol/L | None | >159 umol/L |
| Direct Bilirubin | umol/L | None | >1.35 x ULN |
| Gamma<br>Glutamyl<br>Transferase | U/L | None | >3 x ULN |
| Glucose<br>(fasting) | mmol/L | None | <3 mmol/L<br>>22 mmol/L |
| Magnesium | mmol/L | None | <1 mmol/L<br>>4 mmol/L |
| Phosphorus | mmol/L | None | >0.323 mmol/L above ULN or below LLN |
| Potassium | mmol/L | None | >0.5 mmol/L below LLN<br>>1.0 mmol/L above ULN |
| Sodium | mmol/L | None | >5 mmol/L above ULN or below LLN |
| Total Bilirubin | umol/L | None | >1.5 x ULN |
| Total Protein | g/L | None | >15 g/L above ULN or below LLN |
| Uric acid | umol/L | None | >654 umol/L |
| Free Fatty Acids | mmol/L | None | None |
| HDL Cholesterol | mmol/L | None | None |
| LDL Cholesterol | mmol/L | None | None |
| Triglycerides | mmol/L | None | > 9.04 mmol/L |
| Total<br>Cholesterol | mmol/L | None | None |

204682

| Liver Function Tests | |
|----------------------|-----------------------------------------|
| Laboratory Test | Potential Clinical Concern Value |
| ALT | ≥2 x ULN |
| | ≥ 3 x ULN |
| | ≥ 5 x ULN |
| | ≥8 x ULN |
| | ≥ 10 x ULN |
| | ≥ 3 x ULN and Total Bilirubin ≥ 2 x ULN |
| AST | ≥2 x ULN |
| | ≥ 3 x ULN |
| | ≥ 5 x ULN |
| | ≥8 x ULN |
| | ≥ 10 x ULN |
| | ≥ 3 x ULN and Total Bilirubin ≥ 2 x ULN |
| Total Bilirubin | ≥ 1.5 x ULN |
| | ≥ 2 x ULN |
| | ≥ 3 x ULN |
| | ≥ 5 x ULN |
| | ≥8 x ULN |
| | ≥ 10 x ULN |

204682

# 10.4. Appendix 4 – Abbreviations & Trade Marks

# **Abbreviations**

| ADA | American Diabetes Association |
|------------|--------------------------------------------------------|
| AE | adverse event |
| ALT (SGPT) | alanine aminotransferase (serum glutamic pyruvic |
| | transaminase) |
| AST (SGOT) | aspartate aminotransferase (serum glutamic oxaloacetic |
| | transaminase) |
| BMI | body mass index |
| BUN | blood urea nitrogen |
| CI | confidence interval |
| CONSORT | Consolidated Standards of Reporting Trials |
| CPK | creatine phosphokinase |
| CV | cardiovascular |
| DCC | dual chamber cartridge |
| DNA | deoxyribonucleic acid |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| eGFR | estimated glomerular filtration rate |
| ELISA | enzyme-linked immunosorbent assay |
| EMA | European Medicines Agency |
| FDA | US Food and Drug Administration |
| FFA | free fatty acids |
| FPG | fasting plasma glucose |
| FRP | females of reproductive potential |
| FSH | follicle stimulating hormone |
| GCP | Good Clinical Practice |
| GCSP | Global Clinical Safety and Pharmacovigilance |
| GGT | gamma glutamyl transferase |
| GI | gastrointestinal |
| GLP-1 | glucagon-like peptide-1 |
| GSK | GlaxoSmithKline |
| HA | human albumin |
| HbA1c | glycated hemoglobin |
| HBcAb | hepatitis B core antibody |
| HBsAg | hepatitis B surface antigen |
| HIV | human immunodeficiency virus |
| hCG | human chorionic gonadotrophin |
| HDL-c | high density lipoproteins |
| HRP | horseradish peroxidase |
| HRT | hormone replacement therapy |

204682

| | 204682 |
|---------------------|-------------------------------------------------------|
| IB | Investigator's Brochure |
| ICH | International Conference on Harmonization |
| IEC | Independent Ethics Committee |
| INR | international normal range |
| IP | investigational product |
| IRB | Institutional Review Board |
| ISRs | injection site reactions |
| ITT | intent-to-treat |
| IVRS | Interactive Voice Response System |
| LDH | lactate dehydrogenase |
| LDL-c | low density lipoproteins; |
| LMCF | last mean carried forward |
| K <sub>2</sub> EDTA | di-potassium ethylenediaminetetraacetic acid |
| MACE | major adverse cardiovascular event |
| MCH | mean corpuscular hemoglobin |
| MCV | mean corpuscular volume |
| MDRD | Modification of Diet in Renal Disease |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MEN-2 | multiple endocrine neoplasia type 2 |
| MI | myocardial infarction |
| MSDS | Material Safety Data Sheet |
| MTC | medullary thyroid cancer |
| OC RDC | Oracle Clinical Remote Data Capture |
| PAC | Pancreatitis Adjudication Committee |
| PD | pharmacodynamics |
| PK | pharmacokinetics |
| PP | per protocol |
| PTS-DPMK | Platform Technologies and Science-Drug Metabolism and |
| | Pharmacokinetics |
| RAP | Reporting Analysis Plan |
| RBC | red blood cell |
| RNA | ribonucleic acid |
| s.c. | subcutaneous |
| SAC | Statistical Analysis Complete |
| SAE | serious adverse event |
| SmPC | Summary of Product Characteristics |
| SRM | Study Reference Manual |
| SU | sulfonylureas |
| T2DM | type 2 diabetes mellitus |
| TSH | thyroid stimulating hormone |
| ULN | upper limit of normal range |
| WBC | white blood cell |
| WCBP | women of child bearing potential |

204682

# **Trademark Information**

Trademarks of the GlaxoSmithKline group of companies

NONE

Trademarks not owned by the GlaxoSmithKline group of companies

MedDRA

204682

# 10.5. Appendix 5: List of Data Displays

# 10.5.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Listings | Tables |
|------------------|----------|--------|
| Study Population | 1 to 4 | 1 |
| Safety | 5 to 17 | |

# 10.5.2. Study Population Tables

| Stud | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No | Popula<br>tion | IDSL /<br>TST ID /<br>Exampl<br>e Shell | Title | Programming Notes | Delivera<br>ble<br>[Priority] |
| [Den | [Demographics and Baseline Characteristics] | | | | |
| 1.1. | [Safety] | | Demographic Characteristics | | |

204682

# 10.5.3. Listings

| Listi | Listings | | | | |
|---|---|---|---|---|---|
| No | Popula<br>tion | IDSL /<br>TST ID /<br>Exampl<br>e Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1. | [Safety] | | Inclusion/Exclusion Criteria Deviations | | |
| 2. | [Safety] | | Demographics and Baseline<br>Characteristics | | |
| 3. | [Safety] | | Geographic Ancestry | | |
| 4. | [Safety] | | Concomitant Medications | | |
| 5. | [Safety] | | Albiglutide Administration | | |
| 6. | [Safety] | | Adverse Events | | |
| 7. | [Safety] | | Hematology Laboratory Evaluations | | |
| 8. | [Safety] | | Chemistry Laboratory Evaluations | | |
| 9. | [Safety] | | Urinalysis Laboratory Evaluations | | |
| 10. | [Safety] | | Laboratory Data for Subjects with Any Value of Potential Clinical Importance | | |
| 11. | [Safety] | | Liver Functions with Any Value of Potential Clinical Importance | | |
| 12. | [Safety] | | Vital Signs | | |
| 13. | [Safety] | | ECG Values | | |
| 14. | [Safety] | | Overall ECG Interpretations | | |
| 15. | [Safety] | | Product Investigator's Comments | | |
| 16. | [Safety] | | Drug Accountability | | |
| 17. | [Safety] | | Immunogenicity Information: Anti-<br>Albiglutide Antibody | | |